CLINICAL TRIAL: NCT01309815
Title: Existential Issues in Elderly People With Cancer in an Early Palliative Phase- a Phenomenological Hermeneutic Approach
Brief Title: Existential Issues in Elderly People With Cancer
Status: Completed | Type: Observational
Sponsor: Sykehuset Innlandet HF (Other)
Responsible Party: Principal Investigator, Sigrid Helene Kjørven Haug, PhD Researcher, Sykehuset Innlandet HF
Other Study IDs: Haug, SKH
Record Dates: First submitted 2011-03-04; First posted 2011-03-07 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Cancer
Keywords: neoplasms; existentialism; existential concerns; Meaning making; early palliative phase; elderly
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cancer in elderly people: other

SUMMARY:
The purpose is to describe, interpret and provide a detailed understanding of what it means to be elderly people with cancer who receive treatment in specialized health care. Focus is especially put on the content and expression of existential issues and the importance of spirituality for the patient´s life story and medical story.

DETAILED DESCRIPTION:
Existential and spiritual issues in elderly people with cancer are scarcely investigated with respect to the content and importance of these aspects to this patient group in terms of living with their disease and benefit from specialist health treatment and care. The present study is an independent doctoral study that also has an initial function for an intended multidisciplinary research project with the working title "Aged people with cancer".

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer from the age 70 and older receiving palliative treatment in specialized health care

Exclusion Criteria:

* Terminal patients
* Patients considered as too sick for the interview session
* Patients with lack of consent

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Cancer patients from 70 years and older, receiving palliative treatment and care in Innlandet Hospital Trust
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2011-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars J Danbolt, Professor, Principal Investigator — Innlandet Hospital Trust, Centre for Psychology of Religion
Locations (1):
- Innlandet Hospital Trust, Brumunddal, Norway